CLINICAL TRIAL: NCT00339859
Title: DNA Repair, p53 and Apoptosis Phenotypes in Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998027; OH98-C-N027; NCT00559325 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Lung Neoplasms
Keywords: Molecular Epidemiology of Lung Cancer; Health Disparities
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: The population controls are collected from DMV records in the Baltimore region of MD. The cases are patients at the University of Maryland Medical System, including the associated Veterans' Association Hospital.

SUMMARY:
The Laboratory of Human Carcinogenesis and the Pharmocogenetics Section of the Genetic Epidemiology Branch will conduct a lung cancer case-control study in Baltimore, Maryland. The primary hypothesis of the study is to determine if mutagen sensitivity, p53 induction and apoptosis in cultured lymphocytes will be predictive of lung cancer risk. While there are some studies that examine mutagen sensitivity, none of these assays has been well-studied in an epidemiological setting. Because of methodological issues described herein, and the proposed development of new assays, this study will be viewed as a pilot and therefore hypotheses generating. The design of this molecular epidemiology study has been specifically developed to test the reliability and validity of the mutagen sensitivity assay, where a case-control study is needed to assess the possibility of case bias (i.e., results vary due to the concurrent presence of lung cancer rather than risk). Importantly, this protocol will establish a resource that will allow for the validation of these assays and also for the study of other biomarkers and gene-environment interactions, especially those related to DNA repair. Th secondary goals of this study are to 1) demonstrate gene-neuro-behavioral interactions for smoking addiction in controls and 2) assess the relationship of sex-steroid metabolism an and estrogen exposure to lung cancer risk. Cases will have histologically confirmed lung cancer and reside in Baltimore an and surrounding areas. They will be identified through six hospitals in Baltimore. Cases will be recently diagnosed and blood will be collected prior to chemotherapy or radiation therapy. Because of this requirement to obtain samples before treatment (or for surgical cases at least two months after surgery), we recognize that case ascertainment will be reduced, but critical data to assess differences between eligible and ineligible subjects will be collected through tumor registries. Two control groups will be used, the first will be hospital-based (frequency matched by age, gender, race, smoking and hospital) and the second will be population-based (frequency matched by age-, gender and race). The first control group will allow us to examine risk factors for lung cancer independent of smoking (odds ration for smoking = 1.0), and the second will allow the results to be extrapolated to the general population and also will be used to validate the phenotyping assays. The strategy for recruitment will allow us to over-sample for women and African Americans, so that after examination of data for the entire study group, we can assess differences by these subgroups. Cases and controls will receive a structured, in person interview assessing prior medical and cancer history, tobacco use, alcohol use, current medications, occupational history, family medical history, menstrual history and estrogen use, recent nutritional supplements and caffeine intake, and socioeconomic status. The questionnaire also will include the Fagerstrom index for nicotine dependence (FTND), Center for Epidemiologic Studies Depression (CES-D) scale, and a modified version of the Horn-Waingrow Reasons for Smoking (RFS) Scale. The phenotypic markers to be studied will assess DNA repair with cellular response by using lymphocyte cultures exposed in vitro to radiation, bleomycin, benzo(a)pyrene-diol-expoxide and N-methyl-nitrosurea and then measuring induction of chromosomal aberrations, p53 induction and apoptosis. DNA from cases and controls also will be used for genetic polymorphism analysis of carcinogen metabolism, and those relating to the dopaminergic system and nicotinic receptors. Tumors from cases will be evaluated for estrogen and progesterone receptors. The target accrual number of total subjects will be 1,200 where there will be 100 cases for each combination of gender and race (Caucasian- and African Americans), matched to 100 each of the hospital-based and population-based controls.

DETAILED DESCRIPTION:
Background:

The Laboratory of Human Carcinogenesis is conducting an observational non-small cell lung cancer (NSCLC) case-control study in Baltimore, MD. This molecular epidemiology study was developed to test the reliability and validity of the mutagen sensitivity assay, where a case-control study is needed to assess the possibility of case bias. Importantly, this protocol establishes a resource that allows for the study of additional biomarkers and gene-environment interactions. Upon recruitment, cases and controls receive a structured, in person interview assessing prior medical and cancer history, use of tobacco and electronic cigarettes, alcohol use, current medications, occupational history, family medical history, menstrual history and estrogen use, recent nutritional supplements and caffeine intake, and socioeconomic status. Specimen collection consists of a one-time blood sample and/or mouthwash to collect cheek cells (oral cells) and a one-time urine sample. In addition, cancer and surrounding non-cancer tissue that was surgically removed and not needed for diagnosis may be obtained for cases, as well as current medical information from medical records. Primary cell cultures may be established from available fresh tumor tissue. The phenotypic markers to be studied will assess proficiency of DNA repair in lymphocyte cultures exposed in vitro to radiation, bleomycin, benzo(a)pyrene-diol-epoxide by measuring induction of chromosomal aberrations, p53 and apoptosis. DNA from buffy coats or cheek cells will be used for analysis of germline variation in the form of Single Nucleotide Polymorphisms (SNPs) in genes involved in DNA repair, innate immunity, cell cycle control, angiogenesis, apoptosis, cytokines, nicotine addiction, inflammation, hormone metabolism and microRNA. Additionally, IRB approval was received in 2010 to include this study in a multi-institution genome-wide association study (GWAS) of lung cancer in African Americans. Tumors from cases will be evaluated for estrogen and progesterone receptors, somatic mutations, and gene expression. Urine, plasma, serum and tissue sample metabolomics will be analyzed by untargeted approach.

Objectives:

1. To determine if mutagen sensitivity, p53 induction, and apoptosis in cultured lymphocytes are predictive of lung cancer risk.
2. To determine the relationship between sex-steroid metabolism, estrogen exposure, and lung cancer risk.
3. To investigate and develop phenotypic or predictive markers of lung cancer risk and survival, based on mutagen sensitivity, polymorphic markers, gene expression, and metabolomics.
4. To investigate racial disparities associated with lung cancer risk and survival.
5. To examine the relationship between circulating cytokines with risk and survival of lung cancer and to establish the most robust method of cytokine detection.
6. To generate a more accurate measure of ancestry using ancestry informative marker analysis and to integrate this variable into our studies of health disparities
7. To conduct studies of metabolomics on serum, plasma and urine for the purposes of discovering novel markers of risk, diagnosis and prognosis. We will use ultraperformance liquid chromatography coupled to mass spectrometry (UPLS-MS) to search for small molecular weight endogenous metabolites that can classify cancer and predict outcome.

   This is a novel approach for biomarker discovery that also leverages the non-invasive process of biospecimen collection. Tumor and corresponding non tumor tissues from corresponding patients will also be tested using the same methods to extend the discovery of novel tumor metabolites. Further, metabolites of vitamin D will be examined on serum samples from lung cancer cases and controls to assess the relationship between circulating

   levels of Vitamin D metabolites with cancer risk and survival. This analysis will be coupled with testing of Vitamin D pathway SNPs in corresponding patients to determine if certain SNPs are also associated with levels of vitamin D.
8. To evaluate biomarkers of cancer diagnosis and prognosis in circulating tumor DNA
9. To evaluate the microbiome (microbes) present in lung tissue using in situ hybridization of fixed tissues to be completed at Mayo Clinic by collaborators. The collaborators will receive no information on the samples other than their tissue of origin.
10. To collect data and biospecimens on patients that received low dose CT screening as part of their lung cancer diagnosis. This is for the purposes of investigating non-invasive biomarkers of lung cancer diagnosis and prognosis. Low-dose CT screening is now offered at UMMS and the VA for the purposes of early lung cancer detection. These screening guidelines are per CMS guidelines, i.e., age 55-77, >=30 pack-years of smoking and have quit smoking for 15 years or less. Such high-risk patients will be offered annual screening.
11. To culture lung cancer specific microbiome-bacteria from human lung cancers. This work will, in part, be conducted with our collaborator Dr Paul Owrin, who is an expert in the culture of microbial species from human tissues. These samples, approximately 10 per year, will be de-identified of all patient information.
12. To perform RNA analysis of tumor and normal tissues in collaboration with Dr Isidore Rigoustos with the aim of discovering novel signaling pathways in lung cancer.
13. To contribute our data to larger consortia so that we can conduct studies with a higher power and to make valuable, reproducible observations regarding the epidemiology of lung cancer. We will establish this data transfer via a DTA.
14. To conduct next generation DNA sequencing of tumors (and corresponding normal) of patients enrolled in this protocol.
15. To collaborate with intramural colleagues, specifically Dr Jung Byun at NIMHD on the genomic analysis (next generation DNA sequencing) of samples within this contract. We anticipate sending up to 400 samples. No personal identifiable information will be sent or included with these samples.
16. To collaborate with extramural colleagues, specifically Dr John Simmons at Personal Genome Diagnostics, and Dr Peter Campbell at the Welcome Sanger Institute, England, on the genomic analysis (next generation DNA sequencing) of samples within this contract. We anticipate sending up to 400 samples. No personal identifiable information will be sent or included with these samples.
17. To complete MTAs with colleagues outlined in point 16 above.
18. To capture exposures related to reproductive history in both men and women, among both cases and controls and related these exposures to cancer risk and health disparity.
19. To use data collected through the questionnaire to geocode participants.

Eligibility:

* Histologically confirmed NSCLC diagnosed within the past 2 years (case).
* Frequency matched to cases according to age (5-year intervals), gender, and race (population-based control).
* Born in the United States, resident of the state of Maryland
* Subject Characteristics:

  * Speaks English well enough to be interviewed
  * Physically and mentally capable of performing the interview (i.e., must be able to hear the interviewer, mentally comprehend the interviewers questions, and verbally respond)
  * Has never been interviewed as a control for this study
  * Does not currently reside in an institution such as a prison, nursing home, or shelter
  * No history of cancer other than non-melanoma skin cancer or carcinoma in situ of the cervix (population-based control)
  * Has a residential working phone within the home (population-based control)

Design:

* Case/Control; Observational
* Planned statistical analysis: Risk associations between the genotypes and cancer/survival will be assessed using unconditional logistic regression model, with covariate adjustment, as appropriate.
* Number of subjects to be enrolled: Target accrual is 6000 subjects, consisting of 450 cases/each gender in African Americans and 800 cases/each gender in Caucasians. An equal number of controls will be selected for each category of cases based on the combination of gender and race.
* For patients that undergo low dose CT screening at the participating hospitals in this protocol, we will enroll patients that have had a "positive" scan and are attending either UMMS or the VA hospital for further follow up.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Case Subject Selection:

  * Diagnosis of non-small cell lung cancer made pathologically (with confirmation by a second pathologist).
  * Must reside in Baltimore city or contiguous metropolitan counties, Prince George's county or Anne Arundel county.
  * Have a residential working phone within their home.
  * Be born in the United States.
  * Speak English well enough to be interviewed.
  * Be physically and mentally capable of performing the interview (i.e., must be able to hear the interviewer, mentally comprehend the interviewers questions and verbally respond).
  * Never have been interviewed as a control for the study.
  * Consent by the physician from the clinic where the subject was identified, or listed as the treating physician by the tumor registry or surgical pathology report.
  * Report of a positive LDCT screen by a physician
* Hospital-Based Control Selection:

  * Stratified to frequency match cases by age (5 year intervals), gender, race, smoking (20 pack year intervals -- non-smokers, 0-20, 20-40, 40-60 and greater than 60 and ex-smokers [greater than 5 yrs]) and hospital.
  * Must reside in Baltimore city, contiguous metropolitan counties, Prince George's county or Anne Arundel county.
  * Have a residential working phone within their home.
  * Be born in the United States.
  * Speak English well enough to be interviewed.
  * Be physically and mentally capable of performing the interview (i.e., must be able to hear the interviewer, mentally comprehend the interviewers questions and verbally respond).
  * Never have been interviewed as a control for the study.
  * Physician consent by physician from clinic with subject is identified.
* Selection of Population-Based Controls:

  * Stratified to match cases by age (5 year intervals), gender, and race.
  * Must reside in Maryland
  * Have a residential working phone within their home.
  * Be born in the United States.
  * Speak English well enough to be interviewed.
  * Be physically and mentally capable of performing the interview (i.e., must be able to hear the interviewer, mentally comprehend the interviewers' questions and verbally respond).
  * Never been interviewed as a control for the study.

EXCLUSION CRITERIA:

* Case Subject Selection:

  * More than 6 months after initial diagnosis.
  * Currently residing in an institution such as prison, nursing home or shelter.
  * Severely ill in an intensive care unit (after discharge from ICU, then can be reconsidered).
  * Subjects is unable to give informed consent.
* Hospital-Based Control Selection:

  * History of cancer other than non-melanotic skin cancer or in situ cervical cancer.
  * Currently residing in an institution such as a prison, nursing home or shelter.
  * Severely ill in an intensive care unit (after discharge from ICU, the can be reconsidered).
  * Subject is unable to give informed consent.
  * Known diagnosis of HIV, hepatitis B or C.
  * Selection of Population-Based Controls:
  * History of cancer other than non-melanotic skin cancer or in situ cervical cancer.
  * Currently residing in an institution such as a prison, nursing home or shelter.
  * Subjects unable to give informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population controls are collected from DMV records in the Baltimore region of MD. The cases are patients at the University of Maryland Medical System, including the associated Veterans' Association Hospital.@@@
Sampling Method: Non-Probability Sample
Enrollment: 5625 (Actual)
Dates: Start 1995-06-02 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Lung cancer incidence | At diagnosis
  Pathological diagnosis of lung cancer

CONTACTS AND LOCATIONS:
Overall Officials: Brid M Ryan, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Baltimore, Maryland
  - VA Hospital, Baltimore, Baltimore, Maryland